CLINICAL TRIAL: NCT03816345
Title: A Phase Ib Study of Nivolumab in Patients With Autoimmune Disorders and Advanced Malignancies (AIM-NIVO)
Brief Title: Nivolumab in Treating Patients With Autoimmune Disorders and Advanced, Metastatic, or Unresectable Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-00241; NCI-2019-00241 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10204 (Other: University of Texas MD Anderson Cancer Center LAO); 10204 (Other: CTEP); UM1CA186688 (NIH)
Record Dates: First submitted 2019-01-24; First posted 2019-01-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Autoimmune Disease; Crohn Disease; Dermatomyositis; Hematopoietic and Lymphoid Cell Neoplasm; Inflammatory Bowel Disease; Malignant Solid Neoplasm; Multiple Sclerosis; Psoriasis; Psoriatic Arthritis; Rheumatoid Arthritis; Sjogren Syndrome; Systemic Lupus Erythematosus; Systemic Scleroderma; Ulcerative Colitis
MeSH Terms: conditions — Autoimmune Diseases; Crohn Disease; Dermatomyositis; Hematologic Neoplasms; Inflammatory Bowel Diseases; Multiple Sclerosis; Psoriasis; Arthritis, Psoriatic; Arthritis, Rheumatoid; Sjogren's Syndrome; Lupus Erythematosus, Systemic; Scleroderma, Systemic; Colitis, Ulcerative | interventions — Specimen Handling; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood, CSF, tissue, stool, and urine samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood, CSF, tissue, stool and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase Ib trial studies the side effects of nivolumab and to see how well it works in treating patients with autoimmune disorders and cancer that has spread to other places in the body or cannot removed by surgery. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the overall safety, and toxicities associated with the use of the anti-programmed death 1 (PD-1) antibody nivolumab in patients with varying severity of dermatomyositis (DM)/systemic sclerosis (SSc), rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), inflammatory bowel disease (IBD) (ulcerative colitis [UC] and Crohn's disease [CD]), multiple sclerosis (MS), Sjogren's syndrome [SjS], Psoriasis (PsO)/Psoriatic Arthritis (PsA), and other autoimmune diseases.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of nivolumab in terms of objective response rates (ORRs), progression-free survival (PFS), and overall survival (OS) in patients with cancer and DM/SSc, RA, SLE, IBD (UC and CD), MS, SjS, PsO/PsA, and other autoimmune diseases.

II. To observe and record anti-tumor activity. III. To propose dosing recommendations for anti-PD-1 antibodies based on the severity of the autoimmune disorder.

IV. To evaluate the impact of nivolumab on the disease severity indices for: DM/SSc, RA, SLE, IBD: UC and CD, not specified (NS), MS, SjS, PsO/PsA.

V. To identify biomarkers of response and toxicity.

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes every 4 weeks for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo collection of blood, cerebrospinal fluid (CSF), tissue, stool, and urine samples throughout the trial.

After completion of study treatment, patients are followed up for 100 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients can have either histologically confirmed malignancy that is radiologically evaluable and metastatic or unresectable, or have a malignancy for which a PD-1/PD-L1 inhibitor has been approved in the adjuvant setting. Eligible tumor types include solid tumors and malignancies in which there is known evidence of clinical activity for single agent PD-1 or PD-L1 antibodies. Nivolumab is Food and Drug Administration (FDA)-approved for the treatment of melanoma, non-small cell lung cancer (NSCLC), Merkel cell cancer, bladder cancer, renal cell carcinoma (RCC), gastric cancer, hepatocellular carcinoma (HCC), cervical cancer, head and neck cancer, Hodgkin lymphoma (HL), metastatic small cell lung cancer (SCLC), and any solid tumor with microsatellite instability (MSI)-high status confirmed. Patients with HL are eligible but must follow standard response criteria. Additional tumor types may be eligible on a case by case basis upon discussion with principal investigator (PI). Patients enrolling on the trial for adjuvant use will be restricted to those with histology for which a PD-1/PD-L1 inhibitor has been approved in the adjuvant setting including but not limited to NSCLC, melanoma, RCC, cervical cancer, and bladder cancer
* Patients who have previously received other forms of immunotherapy (high-dose [HD] IL-2, IFN, CTLA-4) are allowed. Patients must not have received cytokine immunotherapy for at least 4 weeks before nivolumab administration. Patients who have received prior anti-CTLA4 will be allowed and the washout period is 6 weeks
* Age >= 18 years; children are excluded from this study but may be eligible for future pediatric phase 1 combination trials
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (Karnofsky >= 60)
* Life expectancy of greater than 12 weeks
* Leukocytes >= 1,000/mcL
* Absolute neutrophil count >= 500/mcL
* Platelets >= 50,000/mcL
* Total bilirubin =< 2 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN or =< 8 x institutional ULN for patients with liver metastases or an autoimmune disease that is contributing to the elevation of these values
* Creatinine ULN OR glomerular filtration rate (GFR) >= 30 mL/min (if using the Cockcroft-Gault formula)
* Human immunodeficiency virus (HIV)-infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated
* If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate central nervous system (CNS) specific treatment is not required and is unlikely to be required for at least 4 weeks (or scheduled assessment after the first cycle of treatment), and a risk-benefit analysis (discussion) by the patient and the investigator favors participation in the clinical trial
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab. Women must not be breastfeeding. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception. WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days, and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients with more than one autoimmune disease are eligible. The treating physician would determine which autoimmune disease is dominant and the patient would be treated under that specific cohort

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier have not resolved or stabilized. Palliative (limited-field) radiation therapy (RT) is permitted (2 week washout from start of treatment), if all of the following criteria are met:

  * Repeat imaging demonstrates no new sites of bone metastases
  * The lesion being considered for palliative radiation is not a target lesion
* Patients with prior therapy with an anti-PD-1 or anti-PD-L1
* Patients with prior allogeneic hematologic transplant
* Patients who are receiving any other anticancer investigational agents
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 100 days
  Will be reported overall and by severity, and dose limiting toxicities will be summarized for all patients and by disease severity cohort.
Change in disease assessments | Baseline up to 100 days
  Will be summarized at each time point for each disease severity cohort.
Overall response rate | Up to 100 days
  Will be computed along with its associated exact 95% confidence interval for all patients and by disease severity cohort.
Changes in serum chemokines and circulating immune cells over time | Baseline up to 100 days
  Will be summarized and assessed using generalized linear mixed modeling.
Gene expression in normal tissues | Up to 100 days
  Will be compared with gene expression in malignant tissues based on two-sample t-test and Wilcoxon rank sum test. False discovery rate, if appropriate, will be used to control for multiple testing.
Clinical measures of interest | Up to 100 days
  The association between demographic and clinical measures of interest with overall response rate and toxicity will be evaluated using logistic regression modeling to identify potential predictors of outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Hussein A Tawbi, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (52):
- United States (51):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - HaysMed, Hays, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Cancer Institute Developmental Therapeutics Clinic, Bethesda, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Vaziri H, Turshudzhyan A, Vecchio E. Immunotherapy-induced Colitis: A Comprehensive Review of Epidemiology, Clinical Presentation, Diagnostic Workup, and Management Plan. J Clin Gastroenterol. 2022 Aug 1;56(7):555-564. doi: 10.1097/MCG.0000000000001705. Epub 2022 Apr 21. PMID 35470301